CLINICAL TRIAL: NCT05688306
Title: A Real World Observational Study to Evaluate Thrombosis Risk in Chemotherapy Patients With Solid Tumors Who Receiving Platelet-raising Therapy
Brief Title: To Evaluate Thrombosis Risk in Chemotherapy Patients With Solid Tumors Who Receiving Thrombocytopenia Treatment
Status: Completed | Type: Observational
Sponsor: Liaoning Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Other Study IDs: IL-11xs
Record Dates: First submitted 2022-12-02; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2022-12

CONDITIONS: Chemotherapy-induced Thrombocytopenia
MeSH Terms: interventions — Interleukin-11; Injections; oprelvekin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Recombinant Human Interleukin-11 for Injection — received rhIL-11 injection for at least 5 consecutive days
  Other Names: rhIL-11

SUMMARY:
Chemotherapy-induced thrombocytopenia (CIT) is a common hematological toxicity in patients with solid tumors undergo chemotherapy, which can increase the risk of bleeding, prolong hospital stay, increase medical costs, and even lead to death in severe cases. The incidence and severity of CIT varies among different chemotherapy regimens. Recombinant human interleukin-11 (rhIL-11) and recombinant human thrombopoietin (rhTPO) have been approved for the treatment of chemotherapy-induced thrombocytopenia.

Tumor patients are at high risk for venous thromboembolism (VTE). In the clinical study of rhIL-11, it was found that the administration of rhIL-11 in healthy subjects caused an increase in the plasma concentration of vWF factor in the form of normal mults. The application of rhIL-11 in patients with myeloid leukemia can increase the concentration of α2 globulin, fibrinogen and prothrombin time. However, there have been no large-scale clinical studies at home and abroad to evaluate whether platelet raising therapy will increase the risk of thrombosis in chemotherapy patients with solid tumor. This study is aimed to evaluate the efficacy and safety of platelet upwelling therapy in patients with solid tumors undergoing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathological diagnosis of solid tumors or lymphomas.
* Have received chemotherapy.
* Diagnosed of CIT.
* Continuous use of platelet raising drugs for at least 5 days.

Exclusion Criteria:

* Thrombocytopenia caused other than chemotherapy, including but not limited to: traditional Chinese medicine, congenital platelet disease, etc.
* The basic value of platelet count is continuously higher than 300×10^9/L.
* Those without blood routine or coagulation function data.
* Those who received non-chemotherapy drugs that may cause thrombocytopenia, such as sulfonamides.
* Pseudothrombocytopenia due to Ethylenediamine tetraacetic acid (EDTA) as an anticoagulant in test samples.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with pathological diagnosis of solid tumors or lymphomas
Sampling Method: Non-Probability Sample
Enrollment: 3494 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2022-05-16 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
To assess the incidence of thrombosis. | 1 month after treatment.

SECONDARY OUTCOMES:
To evaluate the absolute count of platelets. | 1 month after treatment.
To evaluate the level D-dimer. | 1 month after treatment.
To examine the coagulation function index. | 1 month after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing Xing, Principal Investigator — Liaoning Cancer Hospital & Institute
Locations (1):
- Xing Xiaojing, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No